CLINICAL TRIAL: NCT01751009
Title: A Randomised Controlled Home-based Trial of the Effects of Fortified Complementary Foods on Vitamin A Status and Body Pool Size in Ghanaian Infants.
Brief Title: Effects of Fortified Complementary Foods on Vitamin A Status and Body Pool Size in Ghanaian Infants.
Acronym: vitapool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kintampo Health Research Centre, Ghana (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IORG0004854
Record Dates: First submitted 2012-11-05; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Malnutrition
Keywords: vitamin A, complementary foods, malnutrition, children
MeSH Terms: conditions — Malnutrition | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin A supplements (Experimental): Sprinkles with Vitamin A
  Interventions: Dietary Supplement: Vitamin A supplements
- Sprinkles without Vitamin A (Active Comparator): Made of other micronutrients without Vitamin A
  Interventions: Dietary Supplement: Sprinkles without Vitamin A

INTERVENTIONS:
Dietary Supplement: Vitamin A supplements — Sprinkles with Vitamin A
  Arms: Vitamin A supplements
Dietary Supplement: Sprinkles without Vitamin A — Active comparator
  Arms: Sprinkles without Vitamin A

SUMMARY:
This study tried to prove that children given food supplements containing vitamin A would have better liver vitamin A stores than children given food supplements without vitamin A over a 5 month period.

DETAILED DESCRIPTION:
The study wanted to assess the effect of fortification of home based complementary foods on vitamin A status in Ghanaian children who receive food supplements known as Sprinkles. The study assessed the vitamin A status and body pool size in children using a test known as the modified relative dose response test (MRDR) tests and stable 13C2 retinol as a tracer, among those who receive Sprinkles with or without vitamin A through home fortification of complementary foods.

ELIGIBILITY:
Inclusion Criteria:

Informed consent of mother of eligible children aged 6-12 months.

Willingness to remain in the study area for entire duration of the study.

Willingness to agree to feed the child with supplied micronutrient supplements for duration of study.

The child should have started taking complementary foods in addition to breast milk.

Child's haemoglobin level of at least 70 g/L.

Exclusion Criteria:

Child's haemoglobin level less than 70 g/L.

Unable to give informed consent

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Vitamin A status after 5 months supplementation | 5 months

SECONDARY OUTCOMES:
acceptability of home based fortified vitamin A supplements | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Tanumihardjo, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Kintampo North Municipality, Kintampo, Ghana

REFERENCES:
- See also: Related Info — http://www.kintampo-hrc.org